CLINICAL TRIAL: NCT01503047
Title: Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tonalin(R)Intake in Overweight People
Brief Title: Conjugated Linoleic Acid (1:1 Isomer Mixture) Intake in Overweight People
Acronym: CLA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Principal Investigator, Ignacio Galicia, Director, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HULP-2297
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CLA group (Experimental): Treatment consisted of exchanging the normal milk product consumed at breakfast for 200 ml of a skimmed milk with a lipid composition of 0.42 g saturated fatty acids (SFAs) and 0.72 g oleic acid, enriched with 3 g of a 1:1 mix of c9-t11 and t10-c12 (Tonalin®) (CLA group)
  Interventions: Dietary Supplement: Tonalin®
- Placebo group (Placebo Comparator): Treatment consisted of exchanging the normal milk product consumed at breakfast for 200 ml of a skimmed milk with a lipid composition of 0.42 g saturated fatty acids (SFAs) and 0.72 g oleic acid, enriched with 3 g oleic acid (placebo, P group.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tonalin® — Treatment consisted of exchanging the normal milk product consumed at breakfast for 200 ml of a skimmed milk with a lipid composition of 0.42 g saturated fatty acids (SFAs) and 0.72 g oleic acid, enriched with 3 g of a 1:1 mix of c9-t11 and t10-c12 (Tonalin®) (CLA group)
  Arms: CLA group
Dietary Supplement: Placebo — Treatment consisted of exchanging the normal milk product consumed at breakfast for 200 ml of a skimmed milk with a lipid composition of 0.42 g saturated fatty acids (SFAs) and 0.72 g oleic acid, enriched with 3 g oleic acid (placebo)
  Arms: Placebo group

SUMMARY:
The aim of the study was to examine the effects and safety of 3 g of a 1:1 mix of c9-t11 and t10-c12 (Tonalin®) on weight control and body composition in healthy overweight individuals who maintained their normal dietary and exercise patterns.

ELIGIBILITY:
Inclusion Criteria:

* aged 30-55 years
* grade II overweight (BMI≥27 but <30 kg/m2)
* not to be adhered to any calorie restriction diet
* not to be taking any weight control medication or have lost more than 5 kg in the three months prior to the study

Exclusion Criteria:

* suffering of serious concomitant disease such as diabetes mellitus type II, metabolic syndrome (according to the criteria of the Adult Treatment Panel III), cancer, kidney disease, HIV, tuberculosis, cardiovascular disease, chronic obstructive pulmonary disease, eating disorders.
* having undergone bariatric surgery and/or intestinal resection
* breastfeeding and pregnancy.
* not to give their signed, informed consent to be included in the study.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
body composition(DXA) | 0, 3, 6 months

SECONDARY OUTCOMES:
anthropometric parameters | 0,1, 2, 3, 4, 5 and 6 month
  paramteres measured were: Weight, Height and Waist Circunference.
Biochemical parameters | 0, 3 and 6 month
  lipid profile glucose, insulin CR-P PAI-1 adiponectin, leptin creatinine GPT and GOT transaminases
HOMA-Index | 0, 3, 6 month
  insulin sensitivity index was calculated using the formula: HOMA-IR = fasting glucose (mmol/l)/fasting immunoreactive insulin (mU/ml)/22•5.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lopez-Plaza B, Bermejo LM, Koester Weber T, Parra P, Serra F, Hernandez M, Palma Milla S, Gomez-Candela C. Effects of milk supplementation with conjugated linoleic acid on weight control and body composition in healthy overweight people. Nutr Hosp. 2013 Nov 1;28(6):2090-8. PMID 24506387
- See also: institution web — http://www.idipaz.es